CLINICAL TRIAL: NCT02634294
Title: Induction of Graft Versus Tumor Effect of Pegylated Interferon Alpha-2b for Patients With Relapsed Hematological Malignancies After Allogeneic Stem Cell Transplantation
Brief Title: Peg Interferon α-2b for Relapsed Hematological Malignancies After Allo-HSCT
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Chun Wang, Director, department of Hematology, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shanghai1st
Record Dates: First submitted 2015-12-05; First posted 2015-12-18 (Estimated); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Hematological Neoplasms; Recurrence
Keywords: Hematological Neoplasms; recurrence; Hematopoietic Stem Cell Transplantation; peginterferon alfa-2b; Graft vs Host Disease
MeSH Terms: conditions — Hematologic Neoplasms; Recurrence; Graft vs Host Disease | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peg interferon alfa-2b (Experimental): Pegylated Interferon α-2b (PEG INTRON®) , 1~1.5μg/kg qw, subcutaneous injection, 1 to 12 months, until occurrence of grade II or higher grade of acute graft versus host disease, or no response to treatment after 8 doses of treatments.
  Interventions: Drug: Peg interferon alfa-2b

INTERVENTIONS:
Drug: Peg interferon alfa-2b — Eligible patients were treated with pegylated interferon alpha-2b (Peg Intron®; Schering-Plough (Brinny) Company, Innishannon, County Cork, Ireland) 1~1.5ug/kg qw, until occurrence of grade II or higher grade of acute graft versus host disease, or no response to treatment after 8 doses of treatments.
  Other Names: PEG INTRON®

SUMMARY:
Aim: to observe the graft versus tumor effect of Pegylated Interferonα-2b in patients with hematological malignancies relapsed after allogeneic hematopoietic stem cell transplantation (alloHSCT) Patients: patients relapsed after alloHSCT, men and women aged 14-60 years, without vital organ dysfunction or ongoing graft-verus-host disease (GVHD).

Number of subjects: 50, Single center, one group, prospective. Drug: pegylated interferon alpha-2b (Peg Intron®; Schering-Plough) 1~1.5ug/kg qw, until occurrence of grade II or higher grade of acute GVHD, or no response to treatment after 8 doses of treatments.

DETAILED DESCRIPTION:
Eligible patients were age 14 to 60 years with molecular, hematological or radiography relapsed hematological malignancies post allogeneic hematopoietic stem cell transplantation.

Molecular relapse was defined as reappearance or 1 log increase of molecular markers or decreasing donor chimerism by more than 5%; Hematological relapse was defined as reappearance of blast in bone marrow smear by more than 5%; radiography relapse was defined as enlargement of lymph nodes by more than 25% or infiltration of tumor cells in other sites.

Patients were excluded if they need immunosuppressant treatment for ongoing grade II～IV acute GVHD or moderate to severe chronic GVHD.

Eligible patients were treated with pegylated interferon alpha-2b (Peg Intron®; Schering-Plough (Brinny) Company, Innishannon, County Cork, Ireland) 1~1.5ug/kg qw, until occurrence of grade II or higher grade of acute GVHD, or no response to treatment after 8 doses of treatments. Patients were followed up every week. Physical exams and blood tests including complete blood count (CBC), chemical were performed every week. Disease status evaluation was performed every month.

Number of subjects: 50 Single center, one group, prospective.

ELIGIBILITY:
Inclusion Criteria:

1. Age 14-60 years, male or female
2. Allo-HSCT recipients with malignant hematological diseases
3. Disease relapse after allo-HSCT, including hematological relapse, molecular relapse
4. Able to provide written informed consent and to comply with all study procedures

Exclusion Criteria:

1. Pregnant or nursing woman
2. Cardiac ejection factor < normal lower limit
3. Active acute or chronic GVHD with immunosuppressant treatment
4. Known hypersensitivity or allergy to interferon
5. Patient might develop serious complications according to investigator's experiences
6. Patient is undergoing other experimental medication

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
response rate of Peg interferon alpha-2b | 90 days
  the percentage of patients acquiring complete remission and partial remission to Peg interferon alpha-2b in 90 days after treatment

SECONDARY OUTCOMES:
overall survival after relapsing | one year
  the percentage of patients still alive after 1 year
disease free survival after relapsing | one year
  the percentage of patients still alive and disease free after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Chun Wang, M.D., Ph.D., Principal Investigator — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Shanghai Jiao Tong University Affilated First People's Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant date available before publication

REFERENCES:
- [Background] Gupta S, Jen J, Kolz K, Cutler D. Dose selection and population pharmacokinetics of PEG-Intron in patients with chronic myelogenous leukaemia. Br J Clin Pharmacol. 2007 Mar;63(3):292-9. doi: 10.1111/j.1365-2125.2006.02757.x. Epub 2006 Aug 30. PMID 16939523
- [Background] Bejanyan N, Weisdorf DJ, Logan BR, Wang HL, Devine SM, de Lima M, Bunjes DW, Zhang MJ. Survival of patients with acute myeloid leukemia relapsing after allogeneic hematopoietic cell transplantation: a center for international blood and marrow transplant research study. Biol Blood Marrow Transplant. 2015 Mar;21(3):454-9. doi: 10.1016/j.bbmt.2014.11.007. Epub 2014 Nov 15. PMID 25460355